CLINICAL TRIAL: NCT01475045
Title: Multicenter, Prospective, Non Interventional Observational Study in Treatments of Asthma and Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: ANASA (Patients' Satisfaction With Pulmonary Diseases' Treatment)
Acronym: ANASA
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 20109-HAL-EL-02; Sponsor ID (Other: Elpen Pharmaceutical Co Inc)
Record Dates: First submitted 2011-10-12; First posted 2011-11-21 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Turbuhaler inhaler use
- Discus inhaler use
- Elpenhaler inhaler use

SUMMARY:
The aim of the study is to compare patients' satisfaction from the use of three different inhalation devices by using the FSI-10 questionnaire

DETAILED DESCRIPTION:
Patients are requested to reply to FSI-10 questionnaire regarding their satisfaction from inhalation devices. Patients are on 3 different asthma inhalation devices with combination treatment (Turbuhaler, Diskus, Elpenhaler)

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old, both genders who are on their inhalation treatment at least two months before study enrollment,
* Who are able to be compliant to study procedures

Exclusion Criteria:

* Patients < 18 years old,
* Patients who are on their inhalation treatment less than two months before study enrollment
* Patients who are not able to be compliant to study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three subgroups of patients who are already in their inhalation treatment (devices: Discus, Elpenhaler, Turbuhaler) are asked to complete the FSI-10 questionnaire valid in Greek language. The questionnaire responses indicate their satisfaction by their treatment devices.
Sampling Method: Probability Sample
Enrollment: 1160 (Actual)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Patients' satisfaction | all study period (5 months)
  Patients' replies to FSI-10 questionnaire valid in Greek language

SECONDARY OUTCOMES:
Patients devices' use | all study period (5 months)

CONTACTS AND LOCATIONS:
Overall Officials: Asimina Gaga, Principal Investigator — 7th Pulmonary Clinic, Sotiria Hospital of Athens
Locations (2):
- Greece (2):
  - 7th Pulmonary Clinic, Sotiria Hospital, Athens
  - Sotiria Hospital, Athens

REFERENCES:
- See also: study design presented in European Respiratory Congress (2 thematric posters) — http://www.erscongress2011.org
- See also: FSI-10 questionnaire has been translated and is valid in Greek language (full article) — http://www.mednet.gr/archives/